CLINICAL TRIAL: NCT00005724
Title: CVD Nutrition Modules Tailored to Low Literacy Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4933; R01HL046775 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Minimal Intervention Group (Other): Pamphlets on healthy eating mailed to participants.
  Interventions: Other: Minimal Intervention Group
- Health Counselor Intervention Group (Experimental): Food for Heart program, a structured diet treatment program for low-income patients with high cholesterol, given by health counselor at 4 treatment visits.
  Interventions: Behavioral: Health Counselor Intervention Group
- Computer Program Intervention Group (Experimental): User-friendly interactive computer program providing dietary counseling tailored to the needs of the participant.
  Interventions: Behavioral: Computer Program Intervention Group

INTERVENTIONS:
Behavioral: Computer Program Intervention Group — A user-friendly, interactive computer program providing dietary counseling tailored to the needs of the participant.
  Arms: Computer Program Intervention Group
Other: Minimal Intervention Group — Dietary Information pamphlets.
  Arms: Minimal Intervention Group
Behavioral: Health Counselor Intervention Group — Food for Heart Program - a structured diet treatment program for low income patients with high cholesterol, given by a health counselor at 4 treatment visits.
  Arms: Health Counselor Intervention Group

SUMMARY:
To develop cardiovascular disease nutrition modules tailored to subjects with low literacy skills.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of an NHLBI initiative on "CVD Nutrition Education for Low Literacy Skills". The initiative originated within the Prevention and Demonstration Branch of the DECA, was approved by the September 1988 National Heart, Lung, and Blood Advisory Council, and released in July 1990.

DESIGN NARRATIVE:

The study had three phases. The goal of Phase I was to develop two innovative care modules that used demographic, psycho-social, nutritional, and behavioral information to individually tailor nutrition treatment programs for southern patients with less than ninth grade reading skills. Counselor Directed innovative care consisted of a structured assessment and intervention package of simply written, graphically-oriented printed materials to guide the patient and health counselor (nutritionist, health educator, nurse, or physician). Computer Assisted innovative care used a user-friendly, interactive, computer assisted program permitting more sophisticated tailoring to individual needs, conveying nutrition information in a vivid, understandable format, and extending the services of the health counselor. The investigators used focus groups of patients with low literacy skills to aid in concept development and refinement of intervention delivery strategies. Reliable and valid assessments of readability and comprehension helped further refine the materials.

In Phase II, a randomized trial was conducted to determine if the innovative modules produced a meaningful reduction in cholesterol and overall cardiovascular risk compared to standard care. Subjects with high cholesterol and low literacy skills served by four community health centers were randomly assigned to one of four groups: Innovative Care-Counselor Directed, Innovative Care-Computer Assisted, Standard Care, and Usual Care for dietary treatment of cholesterol, obesity, and hypertension. Standard Care involved the same amount of time and health counselor exposure as Innovative Care, but used currently available materials. Usual Care patients were referred to their usual provider for treatment. After four months and again at one year, changes in lipids, blood pressure, and weight were assessed..

Phase Ill consisted of a feasibility study to test the ability of both innovative care modules to reach low literacy adults through county health departments, worksites, and churches. Results of the feasibility assessment helped refine a dissemination strategy using the state health department as a centralized coordinating agency, and county health departments to implement the interventions at the community level.

ELIGIBILITY:
Must have high cholesterol; Low-literacy skills; Must be patient at one of 9 community health centers recruited for study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 1991-08 (Actual); Primary Completion 1995-07 (Actual); Study Completion 1996-07-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 3-month follow-up
  Total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Keyserling, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No